CLINICAL TRIAL: NCT01782339
Title: A Novel Single Arm Phase II Study for Relapsed Germ Cell Tumours With Poor Prognosis
Acronym: GAMMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007755; 2010-022795-31 (EudraCT Number)
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Germ Cell Tumour
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Drug Therapy, Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Chemotherapy (Experimental): 4 cycles of: Day 1 Actinomycin D 1mg/m2, Paclitaxel 80mg/m2, Methotrexate Day 4 Oxaliplatin 100mg/m2 Pegfilgrastim 6mg Day 8* Paclitaxel 80mg/m2 Day 15 Paclitaxel 80mg/m2
  *Day 8 will be omitted for the first three patients treated in this study and will be given at the end of treatment in a fifth cycle where Paclitaxel 80mg/m2 will be administered on Days 1, 8, 15 and 22. Before adding the extra Paclitaxel 80mg/m2 dose on day 8 the safety data for these patients will be reviewed by a DMC.
  NB This 5th cycle for patients 1-3 has been included to ensure that the four 'missed doses of paclitaxel are not omitted from the patients treatment regimen. Cycles 1-4 are 21 days cycles; Cycle 5 (for the first three patients only) is a 28 day cycle.
  Interventions: Drug: Combination Chemotherapy

INTERVENTIONS:
Drug: Combination Chemotherapy — 4 cycles of: Day 1 Actinomycin D 1mg/m2, Paclitaxel 80mg/m2, Methotrexate Day 4 Oxaliplatin 100mg/m2 Pegfilgrastim 6mg Day 8* Paclitaxel 80mg/m2 Day 15 Paclitaxel 80mg/m2
  *Day 8 will be omitted for the first three patients treated in this study and will be given at the end of treatment in a fifth cycle where Paclitaxel 80mg/m2 will be administered on Days 1, 8, 15 and 22. Before adding the extra Paclitaxel 80mg/m2 dose on day 8 the safety data for these patients will be reviewed by a DMC.
  NB This 5th cycle for patients 1-3 has been included to ensure that the four 'missed doses of paclitaxel are not omitted from the patients treatment regimen. Cycles 1-4 are 21 days cycles; Cycle 5 (for the first three patients only) is a 28 day cycle.

SUMMARY:
The treatment of germ cell tumours is considered to be one of the major successes in the area of cytotoxic chemotherapy. Even in patients who relapse after first line therapy, a durable remission rate of between 25% and 60% has been seen using further chemotherapy. In 1999, researchers at St Bartholomew's Hospital developed the GAMEC protocol (combination chemotherapy with filgrastim, actinomycin D, methotrexate, etoposide, cisplatin). Results from this study showed that 50% of patients with relapsed testicular cancer could be cured using this treatment. When we reviewed the individual patients it was clear that older patients (>35yrs) or patients with a raised Lactate Dehydrogenase (a blood test that monitors cancer activity), did not do as well. In addition, patients whose original tumour started in their chest (mediastinal germ cell tumour) have tended to do badly if they relapse. We have been developing a study for patients who fulfil at least one of these criteria. The GAMIO study (filgrastim, actinomycin D, methotrexate, irinotecan, oxaliplatin) has recently closed due to problems with high levels of toxicity from the irinotecan. GAMMA is a new study that will use paclitaxel instead of irinotecan and oxaliplatin instead of cisplatin. We expect that this treatment with oxaliplatin will be less damaging to the kidneys than cisplatin. Both oxaliplatin and paclitaxel and oxaliplatin and irinotecan have similar activity in relapsed patients in the phase II setting. We hope to improve on our previous results with this substitution and see if this will lead to an improvement in the cure rate of relapsed germ cell tumours with poor prognosis and reduce the side effects compared to our standard treatment. In addition, we do not expect any hearing damage and the treatment requires a shorter hospital stay.

DETAILED DESCRIPTION:
Patients will receive a 4 drug combination chemotherapy in hospital over two nights. On the third day, the patient will receive an injection of pegfilgrastim. This stimulates the bone marrow to produce white blood cells and shortens the period of risk of serious infection. The treatment will be repeated every three weeks. This constitutes one cycle of treatment. We aim to give the patient four cycles of treatment over a total of twelve weeks.

Before each cycle, the following will be conducted - physical examination, full blood count, urea + electrolytes, liver function tests, LDH, αFP, βHCG.

Patients will have a FDG PET-CT scan at baseline, prior to cycle 2(approximately 1521 days after chemotherapy starts)and within 28 days of the last treatment, only if clinically indicated. On each cycle, serum creatinine should be measured 24 hours after the start of the methotrexate to exclude renal failure due to methotrexate.

The following will be conducted at the end of treatment physical examination, full blood count, urea + electrolytes, liver function tests, LDH, αFP, βHCG. The patients will be monitored during chemotherapy and then monthly in the first year and two monthly in the second year.

An interim analysis will be performed after 15 patients have completed treatment. If less than 9 responses are observed in this group, the study will be terminated. The final analysis will be performed after 43 patients have recruited, completed treatment and been followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Germ Cell Tumour (GCT)
* Relapsed or progression on or following platinum-based chemotherapy (rising tumour markers or progressive disease on PET CT Scan prior to entering study)
* Neutrophil count >1.0x109/l
* Platelets >70x109/l
* Haemoglobin >100g/l (may be transfused)
* Glomerular filtration rate >40ml/min (determined by EDTA clearance or calculated creatinine clearance using the Cockcroft - Gault equation if unable to perform EDTA clearance)
* Males and females aged 16-65 years

  a) Male patients must have IGCCCG2 prognostic score, low to very high
* Patients must be sterile or agree to use adequate contraception during the period of therapy
* ECOG Performance status 0-3
* Able and willing to give written informed consent and comply with the protocol study procedures.

Exclusion Criteria:

* Other malignancy except basal cell carcinoma
* Significant co-morbidity likely to make delivery of this treatment unsafe
* Currently enrolled in any other investigational drug study
* Previous chemotherapy with oxaliplatin, methotrexate or Actinomycin D
* Patients who have peripheral neuropathy with functional impairment

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2 years

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
Overall Survival | 2 years
Toxicity Level | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dr Shamash, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Background] Bedano PM, Brames MJ, Williams SD, Juliar BE, Einhorn LH. Phase II study of cisplatin plus epirubicin salvage chemotherapy in refractory germ cell tumors. J Clin Oncol. 2006 Dec 1;24(34):5403-7. doi: 10.1200/JCO.2006.05.8065. PMID 17135640
- [Background] Haba Y, Williams MV, Neal DE, Ong JY, Ostrowski MJ, Ell PJ, Nargund V, Shamash J, Oliver RT. Stage migration and pilot studies of reduced chemotherapy supported by positron-emission tomography findings suggest new combined strategies for stage 2 nonseminoma germ cell tumour. BJU Int. 2008 Mar;101(5):570-4. doi: 10.1111/j.1464-410X.2007.07387.x. PMID 18257857
- [Background] Pectasides D, Pectasides M, Farmakis D, Aravantinos G, Nikolaou M, Koumpou M, Gaglia A, Kostopoulou V, Mylonakis N, Economopoulos T, Raptis SA. Oxaliplatin and irinotecan plus granulocyte-colony stimulating factor as third-line treatment in relapsed or cisplatin-refractory germ-cell tumor patients: a phase II study. Eur Urol. 2004 Aug;46(2):216-21. doi: 10.1016/j.eururo.2004.03.001. PMID 15245816
- [Background] Shamash J, Powles T, Ansell W, Berney D, Stebbing J, Mutsvangwa K, Wilson P, Asterling S, Liu S, Wyatt P, Joel SP, Oliver RT. GAMEC--a new intensive protocol for untreated poor prognosis and relapsed or refractory germ cell tumours. Br J Cancer. 2007 Aug 6;97(3):308-14. doi: 10.1038/sj.bjc.6603865. Epub 2007 Jul 3. PMID 17609665
- [Background] Shamash J, Powles T, Mutsvangwa K, Wilson P, Ansell W, Walsh E, Berney D, Stebbing J, Oliver T. A phase II study using a topoisomerase I-based approach in patients with multiply relapsed germ-cell tumours. Ann Oncol. 2007 May;18(5):925-30. doi: 10.1093/annonc/mdm002. Epub 2007 Mar 12. PMID 17355956
- [Background] Theodore C, Chevreau C, Yataqhene Y, Fizazi K, Delord JP, Lotz JP, Geoffrois L, Kerbrat P, Bui V, Flechon A. A phase II multicenter study of oxaliplatin in combination with paclitaxel in poor prognosis patients who failed cisplatin-based chemotherapy for germ-cell tumors. Ann Oncol. 2008 Aug;19(8):1465-1469. doi: 10.1093/annonc/mdn122. Epub 2008 Apr 2. PMID 18385203
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Gerlinger M, Wilson P, Powles T, Shamash J. Elevated LDH predicts poor outcome of recurrent germ cell tumours treated with dose dense chemotherapy. Eur J Cancer. 2010 Nov;46(16):2913-8. doi: 10.1016/j.ejca.2010.07.004. Epub 2010 Aug 13. PMID 20709529
- [Background] International Prognostic Factors Study Group; Lorch A, Beyer J, Bascoul-Mollevi C, Kramar A, Einhorn LH, Necchi A, Massard C, De Giorgi U, Flechon A, Margolin KA, Lotz JP, Germa Lluch JR, Powles T, Kollmannsberger CK. Prognostic factors in patients with metastatic germ cell tumors who experienced treatment failure with cisplatin-based first-line chemotherapy. J Clin Oncol. 2010 Nov 20;28(33):4906-11. doi: 10.1200/JCO.2009.26.8128. Epub 2010 Oct 18. PMID 20956623
- See also: Related Info — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-022795-31/results